CLINICAL TRIAL: NCT07054073
Title: HCMR Re-Imaging Study
Status: Not yet recruiting | Type: Observational
Sponsor: Christopher Kramer (Other)
Collaborators: Brigham and Women's Hospital (Other); Mayo Clinic (Other); Tufts Medical Center (Other); Northwestern University (Other); University of Michigan (Other); The Cleveland Clinic (Other); University Hospital Birmingham NHS Foundation Trust (Other); Glenfield Hospital, Leicester (Other); London Chest Hospital (Unknown); Cytokinetics (Industry); Toronto General Hospital (Other)
Responsible Party: Sponsor-Investigator, Christopher Kramer, University of Virginia Health System, University of Virginia
Organization: University of Virginia (Other)
Other Study IDs: 302244
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Hypertrophic Cardiomyopathy (HCM)
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obstructive HCM
  Interventions: Other: None - observational study
- Non-obstructive HCM
  Interventions: Other: None - observational study

INTERVENTIONS:
Other: None - observational study — None - observational study

SUMMARY:
This study aims to learn what might predict heart problems (like sudden death from a fast heart rhythm or heart failure) in people with a genetic condition called hypertrophic cardiomyopathy (HCM). HCM causes the heart muscle to become thick, which can make the heart stiff and harder to work properly. It can also affect the heart's electrical system.

This study is looking to enroll patients that were previously part of a research project called "HCMR - Novel Predictors of Outcome in Hypertrophic Cardiomyopathy." The results of that study are still being reviewed, but they might show that people who had a substance called Gadolinium (MRI contrast or dye) collected in their heart muscle may have a higher risk for heart problems, including sudden cardiac death. This is called "late gadolinium enhancement" (LGE). This study is aiming to do follow-up imaging on those patients to better understand how LGE affects people with HCM.

ELIGIBILITY:
Inclusion Criteria:

Patients in the original HCMR cohort with:

1. Obstructive HCM

   * Males and females between 18 and 65 years of age
   * BMI < 35 kg/m2
   * LVOT-G at entry as follows:

   Resting gradient ≥50 mmHg OR Resting gradient ≥30 mmHg and <50 mmHg with post-Valsalva LVOT-G ≥50 mmHg

   • NYHA Class II or III or
2. Non-obstructive HCM

   * Same criteria as above except resting LVOT-G is <30mmHg and post-Valsalva gradient <50mm Hg
   * BMI <40kg/m2
   * Elevated NT-proBNP > 300 pg/mL at the time of enrollment
   * LVEF ≥55%

Exclusion Criteria:

* Paroxysmal atrial fibrillation or flutter documented prior to entry.
* Paroxysmal or permanent atrial fibrillation requiring rhythm restoring treatment (eg, direct-current cardioversion, ablation procedure, or antiarrhythmic therapy) ≤6 months prior to entry. (This exclusion does not apply if atrial fibrillation has been treated with anticoagulation and adequately rate-controlled for >6 months.)
* History of syncope or sustained ventricular tachyarrhythmia with exercise within 6 months prior to entry.
* Pregnancy due to potential risk of gadolinium to the fetus
* Patients with a pacemaker that are pacer-dependent as they cannot undergo MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants from the HCMR original cohort who also meet this study's eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in % LGE mass | From baseline over a minimum of 7 years
  To assess the change in LGE extent from baseline over a minimum of 7 years of follow-up extent in HCM patients who would have been candidates for clinical trials of aficamten.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kramer, MD, Principal Investigator — University of Virginia; Stefan Neubauer, MD, Principal Investigator — University of Oxford
Locations (8):
- United States (6):
  - Northwestern, Evanston, Illinois
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Tufts Medical Center, Medford, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Cleveland Clinic, Cleveland, Ohio
  - University of Virginia, Charlottesville, Virginia
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - London Chest Hospital, London

DOCUMENTS (2):
  • Study Protocol (2025-02-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT07054073/Prot_000.pdf
  • Informed Consent Form (2025-02-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT07054073/ICF_001.pdf